CLINICAL TRIAL: NCT06176053
Title: Feasibility and Acceptability of Home-based Stretching Exercises in Patients With Fibromyalgia
Brief Title: Feasibility and Acceptability of Home-based Stretching Exercises in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College of Northern Denmark (Other)
Collaborators: Bispebjerg Hospital (Other); University of Copenhagen (Other); Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Feasibility and acceptability
Record Dates: First submitted 2023-12-08; First posted 2023-12-19 (Actual); Last update posted 2024-06-28 (Actual); Status verified 2024-06

CONDITIONS: Fibromyalgia; Pain; Quality of Life
MeSH Terms: conditions — Fibromyalgia; Pain

STUDY DESIGN:
Intervention Model Description: Feasibility and acceptability study
Masking Description: Participants were blinded to the results of all measurements and naïve to research hypotheses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Regular statict stretching for six weeks (Experimental): Twelve patients aged 18-65, diagnosed with fibromyalgia, will be recruited to participate in a six-week, supervised, home-based stretching program. Exercises are to be performed daily (6 minutes per day) for six weeks. Adherence will be supported, and weekly contact with each participant will be maintained via a mHealth application.
  Interventions: Other: Homebased stretching exercise and app supervision

INTERVENTIONS:
Other: Homebased stretching exercise and app supervision — The intervention group will perform a self-administered, home-based stretching program (a total of 6 minutes per day) and maintain their daily activities as identified at baseline. Exercises are to be performed daily for six weeks. Adherence will be supported, and weekly contact with each participant will be maintained via a mHealth application.

SUMMARY:
The study aims to gather knowledge about the patient's acceptance of the intervention and testing procedures, assess the adherence to the intervention, estimate the recruitment rate, and inform the sample size calculation for a subsequent randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients are included if they are aged 18 to 55 years and diagnosed with fibromyalgia in accordance with the American College of Rheumatology (ACR) criteria

Exclusion Criteria:

* Non-controlled systemic disorders
* Impaired alertness or comprehension
* relevant joint disorders (e.g., severe arthritis, arthroplasty of the hip or knee, and rheumatoid arthritis)
* recent changes in therapy
* neurological and musculoskeletal conditions that could compromise assessments

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Pressure pain thresholds | Pressure pain thresholds were measured as a baseline before the participants are instructed in the home exercises
  Pressure pain thresholds was measures using a handheld pressure algometer
Pressure pain thresholds | Pressure pain thresholds were measured six-weeks after the intervention started
  Pressure pain thresholds was measured using a handheld pressure algometer

SECONDARY OUTCOMES:
Health related Quality of Life | Quality of life was measured as a baseline before the paticipants are instructed in the home exercises
  Quality of life measured by the SF-36 Short Form
Health related Quality of Life | Quality of life was measured six-weeks after the intervention started
  Quality of life measured by the SF-36 Short Form
Range of motion | Range of motion was measured as a baseline before the participants were instructed in the home exercises
  Passive knee extension range of motion measured by the Biodex system 4 pro isokinetic dynamometer
Range of motion | Range of motion was measured six-weeks after the intervention started
  Passive knee extension range of motion measured by the Biodex system 4 pro isokinetic dynamometer

OTHER OUTCOMES:
Fibromyalgia symptoms | Fibromyalgia symptoms were measured as a baseline before the paticipants are instructed in the home exercises
  Fibromyalgia symptoms were measure using the The Revised Fibromyalgia Impact Questionnaire (FIQR)
Fibromyalgia symptoms | Fibromyalgia symptoms was measured six-weeks after the intervention started
  Fibromyalgia symptoms were measure using the The Revised Fibromyalgia Impact Questionnaire (FIQR)

CONTACTS AND LOCATIONS:
Overall Officials: Lise Eckardt, Pt. Msc, Study Director — Department of Physiotherapy, University College of Northern Denmark
Locations (1):
- University College of Northern Denmark, Aalborg, Select, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data is made available upon request.
Supporting Information: Study Protocol
Time Frame: The study protocol will be published.
Access Criteria: The study protocol will be published open access

REFERENCES:
- [Derived] Stove MP, Larsen LL, Magnusson SP, Thomsen JL, Riis A. Exploring the feasibility, acceptability and preliminary efficacy of a Home-Based stretching program for adults with fibromyalgia: a prospective Pre-Post feasibility study. Rheumatol Int. 2025 Aug 11;45(9):191. doi: 10.1007/s00296-025-05921-4. PMID 40788404